CLINICAL TRIAL: NCT05173454
Title: Effect of Breastfeeding Education and Support Provided to Male Partners on Optimal Breastfeeding Practice in Hadiya Zone, Southern Ethiopia: A Cluster-Randomized Controlled Trial
Brief Title: Effect of Breastfeeding Education and Support Provided to Male Partners on Optimal Breastfeeding Practice in Ethiopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jimma University (Other)
Collaborators: Nestlé Foundation (Other)
Responsible Party: Principal Investigator, Mulatu Abageda Anamo, Principal Investigator, Jimma University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: RP 0896/11
Record Dates: First submitted 2021-12-04; First posted 2021-12-30 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Breastfeeding; Breast Fed; Breast Feeding, Exclusive; Breastfed; Breastfeeding, Exclusive
Keywords: optimal breastfeeding practice; male partner; education and support; Ethiopia
MeSH Terms: conditions — Breast Feeding | interventions — Palliative Care

STUDY DESIGN:
Intervention Model Description: The study will have two arms, i.e., intervention and control groups. The intervention group will receive antenatal and postnatal breastfeeding education and support and control group will receive routine care.
Who Masked: Outcomes Assessor
Masking Description: The intervention will be single-blinded. The outcome assessors will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breastfeeding Education and Support (Experimental): The intervention arm will receive antenatal and postnatal breastfeeding education and support intervention for six months starting in their third trimester pregnancy period. The intervention package is comprised of four components: Antenatal breastfeeding education, providing specific take-home print materials, Telephone call counseling and Individual home visit.
  Interventions: Behavioral: Breastfeeding Education and Support
- Usual or routine care (No Intervention): The routine care will be continued in the control group.

INTERVENTIONS:
Behavioral: Breastfeeding Education and Support — The trained village health workers will provide breastfeeding education and support for male partners and mothers in intervention group for the six month period. During intervention trained village health workers will cover antenatal breastfeeding education to raise knowledge, awareness, support, and counseling on benefits of optimal breastfeeding practices and involvement in supporting breastfeeding mothers once at third trimester pregnancy period; Specific take-home print materials will be developed that support optimal breastfeeding practices and will be given for both partners during third trimester pregnancy; Telephone call counselling will be held to the male partners on optimal breastfeeding practices and involvement in supporting breastfeeding mothers at second week and third month postpartum and there will be three home visits during 6th week, 3.5 month and 5th month.
  Arms: Breastfeeding Education and Support

SUMMARY:
Optimal breastfeeding practices are essential for child survival, growth, development, and for the health of mothers. Globally, optimal breastfeeding practices are still low and breastfeeding practices are not optimal in Ethiopia. Male partners have an important but often neglected role in the promotion of breastfeeding practices and currently, male partners are not targeted in breastfeeding education provided by health care providers. The effect of breastfeeding interventions delivered to male partners on optimal breastfeeding has not been studied in the Ethiopian context. It is important to investigate breastfeeding promotion education and support provided to male partners compared to the usual care effective in improving optimal breastfeeding practice in lactating mothers. Therefore, in this study cluster-randomized controlled trials will be conducted to evaluate the effect of breastfeeding education and support provided to male partners on optimal breastfeeding practice in Ethiopia.

DETAILED DESCRIPTION:
Optimal breastfeeding practices are essential for child survival, growth, development, and for the health of mothers. Globally, optimal breastfeeding practices are still low: less than 42% of new-borns begin breastfeeding in the first hour after birth, 41% of infants less than 6 months of age are exclusively breastfed and only 45% of mothers continue breastfeeding for at least two years. It's estimated that 823,000 deaths of children could be prevented every year through optimal breastfeeding practices. However, breastfeeding practices are not optimal in Ethiopia. Male partners have an important but often neglected role in the promotion of breastfeeding practices and currently, participants are not targeted in breastfeeding education provided by health care providers. The effect of breastfeeding interventions delivered to male partners on optimal breastfeeding has not been studied in the Ethiopian context.

The aim of this study is to evaluate the effect of breastfeeding education and support provided to male partners on optimal breastfeeding practice in Hadiya Zone, southern Ethiopia. A cluster-randomized controlled trial will be conducted. The intervention will be provided to the mothers and male partners by trained village health workers . The male partners in the intervention group will receive breastfeeding education and support, but participants in the control group will receive routine care. The breastfeeding education and support intervention package is comprised of four components: 1) Paternal and maternal group education, 2) providing specific take-home print materials, 3) Telephone call counseling and 4) Individual home visit. A total of 408 couples in third trimester pregnancy will be recruited to either the intervention group (204) or a control group (204) from 16 clusters. Clusters will be Kebeles (lowest administrative unit). Randomization will be conducted at the cluster level.Study assessors will be masked. Data analysis will be conducted by STATA version 14.0 using an Intention-To-Treat Approach. Generalized Estimating Equation (GEE) model will be used to determine the effect of the intervention on optimal breastfeeding practice. P values < 0.05 will be used to declare statistical significance. The duration of the intervention is six months.

ELIGIBILITY:
Inclusion Criteria:

* Male partner and mother being in the third trimester of pregnancy
* Male partner and Healthy mother with no underlying disease.
* Male partner and Healthy mother with no pregnancy complication.
* Male partner who live with their wives at home or maintain regular communication with them.
* Partners capable of giving informed consent
* Partners living in the selected cluster with no plans to move away during the intervention period

Exclusion Criteria:

* Mother who experienced a pregnancy loss (miscarriage, still birth, neonatal death) during the follow up period
* Mother had serious medical problems
* Couples who divorced or separated or migrated out of the study area during the intervention
* Mother with twins birth
* Infants admitted to neonatal intensive care units at birth

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 408 (Actual)
Dates: Start 2022-07-14 (Actual); Primary Completion 2023-10-25 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Optimal breastfeeding practice | at 6 months
  Mothers will be asked about infant breastfeeding practice includes early initiation of breastfeeding, breastfeeding frequently (24-h recall), exclusive breastfeeding (24-h recall), intended duration of breastfeeding, pre-lacteal feeding, and feeding colostrum. The infant breastfeeding practice scores will be summed to give a total score that could range between 0 and 6. The infant breastfeeding practice scores will be then classified as Poor (0-2), Medium (3-4), or Good (5-6). When the study participants have scored the highest tertiles (good) of infant breastfeeding practice scores will be considered as optimal breastfeeding practices.

SECONDARY OUTCOMES:
Paternal knowledge, attitude and Supportive practice on optimal breastfeeding | Baseline and at month 6
  Paternal knowledge towards optimal breastfeeding practice will be measured using the breastfeeding knowledge questionnaire after validating it. Paternal attitude towards optimal breastfeeding will be measured using the Iowa Infant Feeding Attitude Scale after validating it. The total score will be calculated out of 85, with a minimum of 17 and a maximum of 85. This scale will help to identify the attitude of the male partner for capturing the favourable attitude (above the mean score) and unfavourable attitude (below the mean score) towards breastfeeding. The supportive practice of male partners in optimal breastfeeding practice will be measured by using a questionnaire which will be coded into Yes or No responses and one mark will be awarded for every correct response (yes), zero will be awarded for every incorrect response (no).Hence, the total number of marks in the supportive practice ranged from 0 to 8.
Maternal breastfeeding self-efficacy | Baseline and at month 6
  Maternal Breastfeeding Self-Efficacy refers to a mother's confidence in her ability to breastfeed her infant and it will be measured using the Breastfeeding Self Efficacy Scale-Short Form developed to assess breastfeeding self-efficacy during postnatal period, a 14-item, self-report instrument and scored in 5-point Likert-type scale.Items are presented positively and summed to produce a total score ranging from 14 to 70, with higher scores indicating higher levels of breastfeeding self-efficacy.
Prevalence of child morbidity | at 6
  Prevalence of child morbidity will be measured based on three morbidities such as diarrhea, fever and acute respiratory illnesses (ARIs). Children with at-least one of the three morbidity during intervention period will be considered
Maternal Perceptions on male partners' breastfeeding Support | Baseline and at month 6
  Male partners' support for breastfeeding will be defined as the physical, emotional and psychosocial support the mother receives from her husband during breastfeeding. Maternal perceptions on husbands' breastfeeding Support will be measured by Postpartum Partner Support Scale, a 25-item self-report instrument designed to assess partner postpartum perceptions of support. Items are rated on a 4-point scale to produce a summative score ranging from 25 to 100, with higher scores indicating higher levels of maternal Perceptions on postpartum-specific partner support.

CONTACTS AND LOCATIONS:
Overall Officials: Mulatu A Anamo, MSc, Principal Investigator — Wachemo University; Tefera B Lema, PhD, Study Director — Jimma University; Mubarek Abera, PhD, Study Director — Jimma University
Locations (1):
- Hadiya Zone, Awasa, Southern Nations, Nationalities, and Peoples' Region, Ethiopia

IPD SHARING:
Plan to Share IPD: Yes
Baseline characteristics, outcome measure and statistical analysis
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Derived] Abageda M, Jena BH, Belachew T. Effect of Male Partner-Targeted Breastfeeding Education and Support Interventions on Optimal Breastfeeding Practices in Central Ethiopia: A Cluster Randomized Controlled Trial. Matern Child Nutr. 2025 Apr;21(2):e13764. doi: 10.1111/mcn.13764. Epub 2024 Nov 18. PMID 39558214
- [Derived] Abageda M, Jena BH, Belachew T. Effectiveness of male partner-targeted breastfeeding education and support interventions on mothers' breastfeeding self-efficacy in central Ethiopia: a cluster-randomized controlled trial. Sci Rep. 2024 Aug 9;14(1):18563. doi: 10.1038/s41598-024-68032-3. PMID 39122804